CLINICAL TRIAL: NCT06009393
Title: A Single-Arm, Open-Label, Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-1918 in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Evaluate the Efficacy and Safety of SHR-1918 in Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1918-202
Record Dates: First submitted 2023-08-15; First posted 2023-08-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1918 (Experimental)
  Interventions: Drug: SHR-1918

INTERVENTIONS:
Drug: SHR-1918 — Three administration

SUMMARY:
This is a single-arm, open-label study to assess the reduction of low-density lipoprotein cholesterol (LDL-C) by SHR-1918 in patients with homozygous familial hypercholesterolemia (HoFH).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of functional HoFH by either genetic or clinical criteria as defined in the protocol
2. LDL-C ≥2.6mmol/L at the screening visit
3. Body weight ≥40 kg
4. Receiving stable lipid-lowering therapy for at least 28 days before enrollment.

Exclusion Criteria:

1. Previously diagnosed type 1 diabetes or poorly controlled type 2 diabetes at screening (HbA1c > 8.5%)
2. eGFR <30ml/min/1.73m2 at the screening visit
3. CK >5times ULN at the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated LDL-C from baseline to week 12 | from baseline to week 12

SECONDARY OUTCOMES:
Change in calculated LDL-C from baseline to week 12 | from baseline to week 12

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng D, Wang L, Pi L, Xu Y, Chen J, Wu Y, Wang N, Chen X, Qi S, Feng S, Cheng G, Lv C, Zhu M, Zhu Y. Anti-ANGPTL3 Antibody SHR-1918 for Homozygous Familial Hypercholesterolemia: A Nonrandomized Clinical Trial. JAMA Cardiol. 2026 Jan 7:e254878. doi: 10.1001/jamacardio.2025.4878. Online ahead of print. PMID 41499141